CLINICAL TRIAL: NCT04387682
Title: Myeloid-derived Suppressor Cells (MDSCs) Detection Before and After Beta-glucan Administration in Oral Squamous Cell Carcinoma Patients
Brief Title: Myeloid-derived Suppressor Cells (MDSCs) in OSCC Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 201701065RIPB
Record Dates: First submitted 2020-05-04; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-04

CONDITIONS: Squamous Cell Carcinoma of the Oral Cavity
Keywords: myeloid-derived suppressor cell (MDSC); oral squamous cell carcinoma (OSCC); whole glucan particle (WGP) β-glucan; flow cytometry; recurrence; prognosis
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence

STUDY DESIGN:
Intervention Model Description: Oral squamous cell carcinoma (OSCC) subject and healthy donors (HDs) subject
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OSCC subjects with β-glucan supplement (Other): Oral squamous cell carcinoma subjects with pre-surgical administration of whole glucan particle β-glucan
  Interventions: Dietary Supplement: β-glucan
- Healthy donors (No Intervention): healthy donors without pre-surgical administration of whole glucan particle β-glucan
- OSCC subjects without β-glucan supplement (No Intervention): Oral squamous cell carcinoma subjects without pre-surgical administration of whole glucan particle β-glucan

INTERVENTIONS:
Dietary Supplement: β-glucan — β-glucan, a biological response regulator, derived from yeast has been known for more than 45 years, and has anti-infective and anti-tumor activities. β-glucan is a molecule with a β-1,3-linked D-glucose backbone and β-1,6-linked side chains. Thus far, at least 4 receptors for β-glucan have been discovered in humans, which are surface antigens associated with macrophages or myeloid precursor cells as complement receptor 3 (CR3; CD11b/CD18, Mac-1, αMβ2 integrin) (Vetvicka et al. 1996; Xia et al. 1999), lactosylceramide (Zimmerman et al. 1998), scavenger receptor (Rice et al. 2002) and dectin-1 (Brown et al. 2003; Taylor et al. 2007; Saijo et al. 2007).
  Arms: OSCC subjects with β-glucan supplement

SUMMARY:
Oral squamous cell carcinoma (OSCC) has the highest annual increase in the rate of death among the top 10 leading cancers in Taiwan. This research aimed to explore whether increased anti-tumor immunity for OSCCs reduces the recurrence rate or improves survival. We first identified CD33+/CD11b+/HLA-DR-/low/CD14+/- as myeloid-derived suppressor cell (MDSC) surface markers by using flow cytometry to compare the MDSC frequency of OSCCs with blood samples from healthy donors (HDs). We then re-confirmed the suppression of T cell proliferation and function achieved by co-culturing with OSCC-educated MDSCs. We subsequently explore whether using particulate β-glucan as a food-grade supplement promotes the human immune system via subversion of immune modulatory MDSCs. Lastly, we correlated clinicopathological parameters with MDSCs and β-glucan administration to examine anti-tumor immunity, and to predict the therapeutic effect and prognosis in OSCC patients..

DETAILED DESCRIPTION:
Oral squamous cell carcinoma (OSCC) has the highest annual increase in the rate of death among the top 10 leading cancers in Taiwan. This research aimed to explore whether increased anti-tumor immunity for OSCCs reduces the recurrence rate or improves survival. We first identified CD33+/CD11b+/HLA-DR-/low/CD14+/- as myeloid-derived suppressor cell (MDSC) surface markers by using flow cytometry to compare the MDSC frequency of OSCCs with blood samples from healthy donors (HDs). We then re-confirmed the suppression of T cell proliferation and function achieved by co-culturing with OSCC-educated MDSCs.

Clinically, we enrolled 100 OSCC patients and 30 HDs to demonstrate a significantly higher MDSC frequency in OSCC candidates than HDs. To determine whether using β-glucan as a food-grade supplement promotes the immune system of OSCC patients, we further allocated OSCC patients with and without pre-surgical administration of whole glucan particle β-glucan to groups II and III, respectively (with group I being the HDs).

We will explore whether using particulate β-glucan as a food-grade supplement promotes the human immune system via subversion of immune modulatory MDSCs. Lastly, we correlated clinicopathological parameters with MDSCs and β-glucan administration to examine anti-tumor immunity, and to predict the therapeutic effect and prognosis in OSCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Oral squamous cell carcinoma (OSCC) subjects without other cancer diagnosis
* healthy donors (HDs)

Exclusion Criteria:

* pregnant woman

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-03-21 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival rate or overall survival rate | 2 years
  This research aimed to explore whether particulate β-glucan as a crucial preoperative adjuvant increasing anti-tumor immunity for OSCCs reduces the recurrence rate or improves survival. Clinically, we enrolled 100 OSCC patients and 30 HDs, and further allocated OSCC patients with and without pre-surgical administration of whole glucan particle β-glucan to groups II and III, respectively (with group I being the HDs). we correlated clinicopathological parameters with MDSCs and β-glucan administration to examine anti-tumor immunity, and to evaluate recurrence-free survival rate or overall survival rate in OSCC patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Jung Cheng, DDS, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Result] Albeituni SH, Ding C, Liu M, Hu X, Luo F, Kloecker G, Bousamra M 2nd, Zhang HG, Yan J. Correction: Yeast-Derived Particulate beta-Glucan Treatment Subverts the Suppression of Myeloid-Derived Suppressor Cells (MDSC) by Inducing Polymorphonuclear MDSC Apoptosis and Monocytic MDSC Differentiation to APC in Cancer. J Immunol. 2016 May 1;196(9):3967. doi: 10.4049/jimmunol.1600346. No abstract available. PMID 27183652
- [Result] Allendorf DJ, Yan J, Ross GD, Hansen RD, Baran JT, Subbarao K, Wang L, Haribabu B. C5a-mediated leukotriene B4-amplified neutrophil chemotaxis is essential in tumor immunotherapy facilitated by anti-tumor monoclonal antibody and beta-glucan. J Immunol. 2005 Jun 1;174(11):7050-6. doi: 10.4049/jimmunol.174.11.7050. PMID 15905548
- [Result] Brown GD, Herre J, Williams DL, Willment JA, Marshall AS, Gordon S. Dectin-1 mediates the biological effects of beta-glucans. J Exp Med. 2003 May 5;197(9):1119-24. doi: 10.1084/jem.20021890. Epub 2003 Apr 28. PMID 12719478
- [Result] Chen WC, Lai CH, Chuang HC, Lin PY, Chen MF. Inflammation-induced myeloid-derived suppressor cells associated with squamous cell carcinoma of the head and neck. Head Neck. 2017 Feb;39(2):347-355. doi: 10.1002/hed.24595. Epub 2016 Oct 3. PMID 27696591
- [Result] Gabrilovich DI, Nagaraj S. Myeloid-derived suppressor cells as regulators of the immune system. Nat Rev Immunol. 2009 Mar;9(3):162-74. doi: 10.1038/nri2506. PMID 19197294
- [Result] Gabrilovich DI, Ostrand-Rosenberg S, Bronte V. Coordinated regulation of myeloid cells by tumours. Nat Rev Immunol. 2012 Mar 22;12(4):253-68. doi: 10.1038/nri3175. PMID 22437938